CLINICAL TRIAL: NCT07164443
Title: A Phase 3 Randomized, Double-blind, Placebo-controlled Study of Pasritamig (JNJ-78278343), a T Cell Redirecting Agent Targeting Human Kallikrein 2, + Best Supportive Care Versus Best Supportive Care for Metastatic Castration-resistant Prostate Cancer
Brief Title: A Study of Pasritamig Versus Placebo in Late Line Metastatic Castration-resistant Prostate Cancer (mCRPC)
Acronym: KLK2-comPAS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 78278343PCR3001; 78278343PCR3001 (Other: Janssen Research & Development, LLC); 2025-520927-26-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2025-09-04; First posted 2025-09-10 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Castration-resistant Prostate Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pasritamig Plus Best Supportive Care (BSC) (Experimental): Participants will receive the step-up doses of pasritamig intravenously (IV) on Cycle 1 Day 1 (C1D1) and C1D8, and target dose of pasritamig IV on C1D15 (Cycle 1 duration is 8 weeks). From C2D1 onwards ( Cycle Duration is 6 week), participants will receive pasritamig target dose IV every 6 weeks. Participants will receive study treatment until confirmed progressive disease, death, intolerable toxicity, withdrawal of consent, or end of the study, whichever occurs first. All participants may receive BSC (defined as palliative external beam radiation, low dose steroids, pain medication, bone sparing agents, and needed palliative procedures) at the discretion of the physician.
  Interventions: Biological: Pasritamig; Drug: Best Supportive Care (BSC)
- Placebo Plus BSC (Placebo Comparator): Participants will receive the step-up doses of placebo IV on C1D1 and C1D8, and target dose of placebo on C1D15. From C2D1 onwards, participants will receive placebo target dose IV every 6 weeks and will receive study treatment until confirmed progressive disease, death, intolerable toxicity, withdrawal of consent, or end of the study, whichever occurs first. All participants may receive BSC at the discretion of the physician.
  Interventions: Other: Placebo; Drug: Best Supportive Care (BSC)

INTERVENTIONS:
Biological: Pasritamig — Pasritamig will be administrated through IV infusion.
  Other Names: JNJ-78278343
  Arms: Pasritamig Plus Best Supportive Care (BSC)
Other: Placebo — Placebo will be administrated through IV infusion.
  Arms: Placebo Plus BSC
Drug: Best Supportive Care (BSC) — BSC will be administered as per physician.

SUMMARY:
The purpose of this study is to evaluate the overall survival (length of time from the start of study to date of death from any cause) for pasritamig (JNJ-78278343) in combination with best supportive care (BSC) as compared to placebo with BSC in participants with metastatic castration-resistant prostate cancer (mCRPC; a stage of cancer that has spread beyond the prostate gland and is no longer responding to hormone therapies).

ELIGIBILITY:
Inclusion Criteria

* Histologically confirmed adenocarcinoma of the prostate
* Metastatic castration-resistant prostate cancer (mCRPC): Disease that is metastatic either to bone, any lymph node, or both without clear evidence of metastasis to visceral organs at the time of screening
* PSA greater than or equal to (>=) 2 nanogram per milliliter (ng/mL) at screening
* In the opinion of the investigator, the next best treatment option is a clinical trial
* Participants should have had all life-prolonging therapies for which they are clinically eligible in the opinion of the investigator and to which they have access. Prior therapies could have been given in any disease setting (not limited to mCRPC). In particular, prior treatment specifications include receipt of the following:

Androgen-receptor pathway inhibitor (ARPI): Must have progressed on at least 1 ARPI and unlikely to benefit from retreatment with another ARPI

Taxanes: Should have received at least 2 previous taxane-based regimens. If a participant has received only 1 taxane regimen, the participant is eligible if:

1. Cabazitaxel is not available
2. The participant's physician deems the participant unsuitable to receive a second taxane regimen due to toxicity risk or prior intolerance Note: a taxane-based regimen consists of at least 2 cycles of a taxane (either as a single agent or in combination with other therapies) administered within the same 2-month period.

Radioligand therapy: Should have been previously treated with at least 1 dose of Prostate-specific membrane antigen (PSMA)-targeted lutetium radioligand therapy (eg, lutetium Lu-177 vipivotide tetraxetan), unless one of the following applies:

1. PSMA-targeted lutetium radioligand therapy is unavailable, not accessible, or not clinically indicated.
2. The participant's physician deems the participant unsuitable to receive PSMA-targeted lutetium radioligand therapy.

Polyadenosine diphosphate-ribose polymerase inhibitors (PARPi): Should have been previously treated with PARPi, if the participant has a known germline or somatic BRCA mutation and treatment is available

* Prior orchiectomy or medical castration (receiving ongoing ADT with a GnRH analog [agonist or antagonist]) prior to the first dose of study treatment and must continue this therapy throughout the treatment phase
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Participants are eligible if they have the following values:

A) eGFR >= 30 milliliters per minute (mL/min) B) Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) less than or equal to (<=) 5 times the Upper Limit of Normal (ULN) C) Serum total bilirubin <= 3 * ULN D) Absolute neutrophil count (ANC) >= 1.0 *10^9/per liter (L) E) Hemoglobin >= 8.0 grams per deciliter (g/dL) F) Platelet count >= 75 * 109/L

Exclusion Criteria

* Venous thromboembolic events within 1 month prior to the first dose of study treatment; uncomplicated (Grade <= 2) deep vein thrombosis is not exclusionary
* Active autoimmune disease within the past 12 months that requires systemic immunosuppressive medications (eg, chronic corticosteroid, methotrexate, or tacrolimus)
* Clinically significant pulmonary compromise, particularly a requirement for supplemental oxygen use (>2 liters per minute (L/min) by nasal cannula) to maintain adequate oxygenation
* Prior or concurrent second malignancy (other than the disease under study) for which natural history or treatment could likely interfere with any study endpoints of safety or the efficacy of the study treatment(s)
* Any of the following within 6 months prior to first dose of study treatment:

A) Myocardial infarction B) Severe or unstable angina C) Clinically significant ventricular arrhythmias D) Congestive heart failure (New York Heart Association class II to IV) E) Transient ischemic attack F) Cerebrovascular accident

- Prior treatment with any CD3-directed therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 663 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2028-05-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to 2 years and 8 months
  OS is defined as the time from randomization to date of death due to any cause.

SECONDARY OUTCOMES:
Radiographic Progression-free Survival (rPFS) | Up to 2 years and 8 months
  rPFS assessed by investigator defined as the time from the date of randomization until the date of radiographic disease progression (based on response evaluation criteria in solid tumors [RECIST] v1.1 and prostate cancer working group 3 [PCWG3] criteria) or death, whichever comes first.
Time to Symptomatic Progression | Up to 2 years and 8 months
  Time to symptomatic progression is defined as time from the date of randomization to the date of any of the following (whichever occurs first): (a) the use of external beam radiation therapy to relieve cancer-related symptoms; (b) the need for tumor-related orthopedic surgical intervention; (c) other cancer-related procedures; (d) cancer-related morbid events; (e) initiation of a new systemic anti-cancer therapy because of cancer symptoms.
Time to Skeletal-Related Event | Up to 2 years and 8 months
  Time to skeletal-related event is defined as the time from the date of randomization to the date of first occurrence of any of the following (whichever occurs first): (a) the use of external beam radiation for skeletal or pelvic symptoms; b) the need for tumor-related orthopedic surgical intervention; (c) the occurrence of new bone fractures (cancer-related); (d) the occurrence of tumor-related spinal cord compression.
Progression-Free Survival (PFS) | Up to 2 years and 8 months
  PFS is defined as the date of randomization to the date of first evidence of radiographic progression, clinical progression, or death from any cause, whichever occurs first.
Time to Prostate Specific Antigen (PSA) Progression | Up to 2 years and 8 months
  Time to PSA progression, defined as the time from randomization to the first date of documented PSA progression per PCWG3 criteria. PSA progression is defined as: after a decline from baseline, PSA increases >= 25 percentage (%) and >= 2 nanograms per milliliter (ng/mL) above the nadir, confirmed by a second value >= 3 weeks later (that is, a confirmed rising trend), or If there is no decline from baseline, PSA increases >= 25 % and >= 2 ng/mL from baseline after 12 weeks.
Time to Pain Progression (TTPP) as Assessed by the Brief Pain Inventory-Short Form (BPI-SF) Item 3 Worst Pain in 24 Hours | Up to 2 years and 8 months
  TTPP is defined as the time from the date of randomization to the date of the first observation of pain progression. Pain progression is defined as an increase of at least 2 points from baseline in the BPI-SF worst pain intensity (item 3) observed at 2 consecutive evaluations >= 3 weeks apart. BPI-SF is an 11-item questionnaire, designed to assess severity and impact of pain on daily functions. Total score range from 0 to 10 with 0 representing "no pain" and 10 representing" pain as bad as you can imagine".
Time to Deterioration in Fatigue as Assessed by the European Organisation For Research And Treatment of Cancer Quality of Life Questionnaire-Core-30 (EORTC QLQ-C30) Fatigue Scale Score | Up to 2 years and 8 months
  Time to deterioration is defined as the time from randomization to the date of the first observation of deterioration in Fatigue. Deterioration in Fatigue is defined as an increase of 10 points on the EORTC QLQ-C30 FA scale observed at 2 consecutive evaluations >= 3 weeks apart. The EORTC QLQ-C30 is a widely used tool for assessing the quality of life of cancer patients in clinical trials. Responses to items 1-28 are rated on a 4-point Likert response scale ranging from 1 "Not at all" to 4 "Very much". Two global health status items are rated on a 7-point numeric rating scale from 1 "Very Poor" to 7 "Excellent". Each subscale of the EORTC QLQ-C30 is scored on a range from 0 to 100. Higher scores indicate worse symptoms or problems.
Number of Participants with Adverse Events (AEs) | Up to 2 years and 8 months
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Number of Participants with Abnormalities in Clinical Laboratory Assessments | Up to 2 years and 8 months
  Participants with abnormalities in clinical laboratory parameters (hematology, clinical chemistry etc.) will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (81):
- United States (27):
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - Colorado Clinical Research, Lakewood, Colorado
  - Bay Pines VA Healthcare System, Bay Pines, Florida
  - Florida Cancer Specialists & Research Institute, Fort Myers, Florida
  - East Jefferson General Hospital, Metairie, Louisiana
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - XCancer Omaha / Urology Cancer Center, Omaha, Nebraska
  - NYU Langone Hospitals, Brooklyn, New York
  - NYU Langone Hospital Long Island, Mineola, New York
  - NYU Langone Health Laura and Isaac Perlmutter Cancer Center, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Compass Oncology, Portland, Oregon
  - Oregon Urology Institute, Springfield, Oregon
  - MidLantic Urology, Bala-Cynwyd, Pennsylvania
  - Keystone Urology Specialists, Lancaster, Pennsylvania
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - Gibbs Cancer Center and Research Institute Pelham, Greer, South Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Gibbs Cancer Center, Spartanburg, South Carolina
  - Tennessee Oncology, Chattanooga, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Urology Clinics of North Texas, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology West Texas, Wichita Falls, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Blue Ridge Cancer Care, Roanoke, Virginia
- Australia (5):
  - Warringal Private Hospital, Heidelberg
  - ICON Cancer Care, Kurralta Park
  - Peter MacCallum Cancer Centre, Melbourne
  - Fiona Stanley Hospital, Murdoch
  - Princess Alexandra Hospital, Woolloongabba
- Belgium (6):
  - AZ Sint-Jan, Bruges
  - Cliniques Universitaires Saint Luc, Brussels
  - AZ Maria Middelares, Ghent
  - Chu Helora Hospital La Louviere Site Jolimont, La Louvière
  - CHC MontLegia, Liège
  - Clinique Saint Pierre, Ottignies
- Brazil (2):
  - Centro de Pesquisa e Ensino em Oncologia de Santa Catarina CEPEN, Florianópolis
  - Associacao Hospitalar Moinhos de Vento, Porto Alegre
- Canada (2):
  - BC Cancer Vancouver, Vancouver, British Columbia
  - CHU de Quebec Universite Laval, Québec, Quebec
- China (4):
  - West China Hospital of Sichuan University, Chengdu
  - Nanjing Drum Tower Hospital, Nanjing
  - Fudan University Shanghai Cancer Center, Shanghai
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
- Germany (3):
  - Urologicum Duisburg, Duisburg
  - Krankenhaus NorthWest, Frankfurt am Main
  - Martini-Klinik am UKE GmbH, Hamburg
- Istituto Clinico Humanitas, Rozzano, Italy
- Japan (10):
  - Kyushu University Hospital, Fukuoka
  - Saitama Medical University International Medical Center, Hidaka
  - Kanazawa University Hospital, Kanazawa
  - Kobe University Hospital, Kobe
  - National Hospital Organization Shikoku Cancer Center, Matsuyama
  - National Hospital Organization Tokyo Medical Center, Meguro Ku
  - Toho University Sakura Medical Center, Sakura
  - Yokohama City University Medical Center, Yokohama
  - Yokohama City University Hospital, Yokohama
  - Yokosuka Kyosai Hospital, Yokosuka
- Netherlands (2):
  - Reinier de Graaf Gasthuis, Delft
  - Tergooi, Hilversum
- Poland (2):
  - IN VIVO Sp. z o.o, Bydgoszcz
  - Narodowy Instytut Onkologii im Marii Sklodowskiej Curie Panstwowy Instytut Badawczy, Warsaw
- Puerto Rico (2):
  - Puerto Rico Medical Research Center, Hato Rey
  - Pan American Center for Oncology Trials LLC, Rio Piedras
- South Korea (3):
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Severance Hospital Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
- Spain (4):
  - Hosp. de Jerez de La Frontera, Jerez de la Frontera
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp Virgen de La Victoria, Málaga
- Taiwan (5):
  - Chang Gung Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District
- United Kingdom (3):
  - University College London Hospitals, London
  - The Christie NHS Foundation Trust Christie Hospital, Manchester
  - Royal Marsden Hospital (Sutton), Sutton

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency